CLINICAL TRIAL: NCT01707953
Title: Efficacy of Midodrine for the Prevention of Orthostatic Hypotension During Early Mobilization After Fast-track Hip Arthroplasty - a Randomized, Placebo Controlled Trial.
Brief Title: Efficacy of Midodrine for the Prevention of Orthostatic Hypotension During Early Mobilization After Fast-track Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Oeivind Jans, M.D, Research Fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RH-4074-OJ1; 2012-002572-13 (EudraCT Number)
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Orthostatic Hypotension; Postoperative Orthostatic Intolerance
MeSH Terms: interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midodrine (Experimental): Midodrine Hydrochloride (5mg) administered as capsule 5 and 23 hours after end of surgery.
  Interventions: Drug: Midodrine
- Placebo (Placebo Comparator): Placebo administered as capsule 5- and 23 hours after end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine — Midodrine 5mg as capsule, administered twice (5 and 23 hours after end of surgery).
  Other Names: Gutron
  Arms: Midodrine
Drug: Placebo — Placebo capsule to mimic midodrine
  Arms: Placebo

SUMMARY:
The aim of this study is to examine the efficacy of 5 mg Midodrine (Gutron) vs. placebo on reducing the incidence of orthostatic hypotension during mobilization 6 h after a total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for primary unilateral hip arthroplasty
* Age >= 18 years
* Able to give informed consent

Exclusion Criteria:

* General anaesthesia for the current procedure
* Digoxin treatment.
* history of renal or hepatic failure
* history of glaucoma
* history chronic urinary retention requiring treatment
* history of orthostatic intolerance / hypotension
* other autonomous nervous system disease
* alcohol or drug abuse
* current malignant disease
* females in the fertile age (possible pregnancy or breast feeding)
* Treatment with anticoagulants
* BMI > 40 kg/m2
* Dementia or cognitive dysfunction (investigators evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Orthostatic hypotension | 6 hours after surgery
  Orthostatic hypotension (OH) during early mobilization 6 hours after end of surgery. OH is classified according to international consensus.

SECONDARY OUTCOMES:
Orthostatic hypotension 24 hours after surgery | 24 hours after end of surgery.
Orthostatic Intolerance | 6 and 24 hours after end of surgery
  Orthostatic intolerance is defined as subjective presyncopal symptoms (dizziness, nausea etc.) during mobilization after surgery
Treatment side effects | 6 and 24 hours after end of surgery
  The following side effects to Midodrine are evaluated:
  * Pruritus
  * Headache
  * Supine hypertension
  * Urinary retention

OTHER OUTCOMES:
Haemodynamic response to mobilization 6 and 24 hours after surgery | 6 and 24 hours after end of surgery
  Haemodynamic response to mobilization (supine, sitting and standing):
  * Response in systolic and diastolic blood pressure
  * Response in heart rate.
  * Response in calculated haemodynamic variables (stroke volume, peripheral resistance)
Heart rate variability | before surgery, 6- and 24 hours after surgery
  Heart rate variability measures including spectral analysis and LF/HF ratio at rest and during mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, Proffessor, Study Chair — Rigshospitalet, Section for Surgical Pathophysiology; Oeivind Jans, M.D., Study Director — Rigshospitalet, Section for Surgical Pathophysiology
Locations (3):
- Denmark (3):
  - Gentofte Hospital, Department of orthopaedic surgery, Hellerup
  - Hvidovre Hospital, Department of orthopaedic surgery, Hvidovre
  - Vejle Sygehus, Department of orthopedic surgery, Vejle